CLINICAL TRIAL: NCT02868437
Title: Effectiveness of Self-cross-linked Hyaluronic Acid Gel in the Prevention of Intrauterine Adhesions After Second Trimester Abortion
Brief Title: Effectiveness of Hyaluronic Acid Gel in the Prevention of Intrauterine Adhesions After Second Trimester Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Collaborators: Bilar Medikal, Turkey (Unknown)
Responsible Party: Principal Investigator, Ozlem Dural, M.D., Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ODural
Record Dates: First submitted 2016-08-10; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Placenta Retained; Uterine Diseases
MeSH Terms: conditions — Placenta, Retained; Uterine Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): The patients who are having curettage for retained product after second trimester abortion will also receive an intervention of intrauterine self-cross-linked hyaluronic acid gel after the procedure
  Interventions: Device: intrauterine self-cross-linked hyaluronic acid gel
- Group 2 (No Intervention): The patients who are having curettage for retained product after second trimester abortion will receive no intervention

INTERVENTIONS:
Device: intrauterine self-cross-linked hyaluronic acid gel — intrauterine self-cross-linked hyaluronic acid gel will apply after curettage for retained product after second trimester abortion
  Arms: Group 1

SUMMARY:
This prospective, randomized, controlled study evaluates the efficacy of self-crosslinked hyaluronic acid gel to prevent the development of de-novo intrauterine adhesions following curettage for retained product after second trimester abortion. One group of participants will underwent curettage plus intrauterine application of self-crosslinked hyaluronic acid gel while the other group will underwent curettage alone (control group).

DETAILED DESCRIPTION:
Intrauterine adhesions are the major long-term complication of curettage for retained products of conception. The risk of adhesion is higher after second trimester abortion. This complication may result in infertility, recurrent miscarriages and irregular periods with dysmenorrhea and pelvic pain.

They have been reported that the intrauterine application of auto-crosslinked hyaluronic acid gel following hysteroscopic adhesiolysis or hysteroscopic surgery significantly reduces the formation of post-operative intrauterine adhesions.

The aim of this prospective, randomized, controlled study is to evaluate the efficacy of self-crosslinked hyaluronic acid gel in the reduction of development of de-novo post-curettage adhesions at 2 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject has curettage for retained product after second trimester abortion

Exclusion Criteria:

* History of curettage or other intrauterine surgery
* History of post-abortion complication or infection

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The presence of de-novo post-curettage adhesions | 2 months
  In 2 months following the curettage, Hysteroscopy will perform to observe of whether there is any intrauterine adhesion

SECONDARY OUTCOMES:
The characteristic of the intrauterine adhesions | 2 months
  If any intrauterine adhesion is detected during the Hysteroscopy, American Fertility Society/American Society for Reproductive Medicine classification of intrauterine adhesions will be used to describe to the characteristic of the intrauterine adhesions

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Dural, M.D., Principal Investigator — Istanbul University School Of Medicine, Department of Obstetrics and Gynecology

REFERENCES:
- [Result] Hooker AB, Lemmers M, Thurkow AL, Heymans MW, Opmeer BC, Brolmann HA, Mol BW, Huirne JA. Systematic review and meta-analysis of intrauterine adhesions after miscarriage: prevalence, risk factors and long-term reproductive outcome. Hum Reprod Update. 2014 Mar-Apr;20(2):262-78. doi: 10.1093/humupd/dmt045. Epub 2013 Sep 29. PMID 24082042
- [Result] Guida M, Acunzo G, Di Spiezio Sardo A, Bifulco G, Piccoli R, Pellicano M, Cerrota G, Cirillo D, Nappi C. Effectiveness of auto-crosslinked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic surgery: a prospective, randomized, controlled study. Hum Reprod. 2004 Jun;19(6):1461-4. doi: 10.1093/humrep/deh238. Epub 2004 Apr 22. PMID 15105384